CLINICAL TRIAL: NCT04596813
Title: CYtosorb Modulation of surgiCal infLammatiON During LVAD insErtion
Brief Title: Role of Cytosorb in Left Ventricular Assist Device Implantation
Acronym: CYCLONE-LVAD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: UMC Utrecht (Other); CytoSorbents, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18IC4535
Record Dates: First submitted 2020-09-23; First posted 2020-10-22 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Heart Failure
Keywords: cardiac surgery; inflammation; cytokines; bypass; artificial heart known as LVAD
MeSH Terms: conditions — Heart Failure; Inflammation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- standard of care (No Intervention)
- standard of care and treatment with the Cytosorb® device (Active Comparator)
  Interventions: Device: CytoSorb 300 mL device

INTERVENTIONS:
Device: CytoSorb 300 mL device — Intra-and postoperative CytoSorb hemoadsorption
  Arms: standard of care and treatment with the Cytosorb® device

SUMMARY:
Mechanical circulatory support, specifically implantable continuous flow left ventricular assist device (CF-LVAD) therapy has been established as a viable treatment for rapidly deteriorating patients suffering from end stage heart failure either as bridge or alternative to heart transplantation. However, a large proportion of these patients experience severe complications in the early postoperative period including right ventricular failure or multi organ failure leading to increased mortality. The leading theory explaining these complications involves exaggerated systemic inflammatory response prior to, during and early after CF-LVAD insertion. Among the cytokines IL-6 appears to play a major role. There is increasing demonstration of the efficacy of a cytokine haemoadsorption (HA) technology in attenuating cytokine response and particularly IL-6 in various inflammatory states and emerging data on the safety of the Cytosorb® device in routine and complex cardiac surgery.

The study team hypothesizes that Cytosorb® treatment is feasible and safe in heart failure patients undergoing LVAD insertion and that it is effective in attenuating IL-6 secretion with benefit in the wider inflammatory and metabolic response to this high-risk surgery.

DETAILED DESCRIPTION:
The principle objectives of this study are:

1. To investigate the efficacy of Cytosorb® treatment in attenuating perioperative changes in IL-6 during CF-LVAD implantation
2. To investigate the feasibility, and safety of Cytosorb® treatment during CF-LVAD implantation.
3. To pilot the effect of Cytosorb® treatment on vasoplegia and organ dysfunction with specific focus on right ventricle failure, liver failure and acute kidney injury (AKI).
4. To establish a collaborative biobank of patient's biological samples to allow extensive characterisation of patient phenotype prior to CF-LVAD implantation and their individual inflammatory and metabolic responses to surgery and perioperative management.

ELIGIBILITY:
Inclusion Criteria:

Adult patients (≥18 years), but ≤70 years; Scheduled for elective LVAD implantation with the use of cardiopulmonary bypass; Written informed consent for participation

Exclusion Criteria:

* Poor spoken and/or written language comprehension
* Declined or missing informed consent
* LVAD implant planned without use of CPB
* Total Artificial Heart implantation
* Planned CPB temperature < 32 °C
* AIDS with a CD4 count of < 200/μL
* Severe thrombocytopenia (PLT <50000
* Application of contrast medium on the day of surgery
* Immunosuppressive therapy or long-term therapy with corticosteroids
* Contraindication to anticoagulation with heparin
* Participation in another clinical intervention trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-09-21 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Increase in plasma IL-6 concentration | from baseline to the time of arrival to intensive care unit (approximately 4 hours).

SECONDARY OUTCOMES:
Changes in IL-6 concentrations at various time points after surgery until ICU discharge | from baseline, 6, 12, 24, 48 and 72 hours after surgery and at ICU discharge, approximately 7 days
Incidence of serious device related adverse events from the time of enrolment through ICU discharge | from the time of enrolment through ICU discharge (approximately 7 days)
Feasibility based on number of patients eligible and receiving study intervention | From Baseline through ICU discharge (approximately 7 days)
  Ratio of eligible patients and those receiving study intervention
Incidence and progression of vasoplegia | from baseline to 24 hours after surgery
  Defined as haemodynamic instability fulfilling the following criteria for at least three consecutive hours during the first 48h after ICU arrival: MAP ≤50 mmHg or SVR ≤800 dynes·s·cm- 5; CI ≥ 2.5 l·min- 1·m- 2; use of norepinephrine ≥200 ng·kg- 1·min- 1 or equivalent doses of vasopressors (epinephrine ≥200 ng·kg- 1·min- 1; dopamine ≥30 μg·kg- 1·min- 1; phenylephrine ≥2 μg·kg- 1·min- 1, or vasopressin ≥0.08 U·min- 1)
Prevalence of right ventricle dysfunction | From baseline to 72 hours after surgery
  Transesophageal echocardiography indices of right ventricle dysfunction based on TAPSE, estimates of the RV-PA coupling, 3D volumetry and ventricle free wall strain
Incidence and progression of Acute Kidney Injury (KDIGO criteria) | From Baseline through ICU discharge (approximately 7 days)
Prevalence of liver dysfunction | from baseline to 72 hours after surgery
  14. Defined as changes in indocyanine green plasma disappearance rate masured by the LiMON® monitor
Sequential Organ Failure Assessment Score (SOFA) | From Baseline through ICU discharge (approximately 7 days)
  Total Daily SOFA Score. The score ranges from 0 (best outcome) to 24 (worst outcome).
Time of mechanical ventilation | From Baseline through ICU discharge (approximately 7 days)
  Duration of invasive mechanical ventilation
Length of ICU stay | From Baseline through ICU discharge (approximately 7 days)
28 day mortality | 28 days after surgery

OTHER OUTCOMES:
Changes in inflammasome analyses | from baseline, 6, 12, 24, 48 and 72 hours after surgery and at ICU discharge, approximately 7 days
  Plasma and urinary levels of the inflammatory mediators: IL-1β,IL-1Ra, IL-6, IL-8, IL-10, TNF-α, MPO and HBP [pg/ml for all]
Changes in the metabolomics profile | from baseline, 6, 12, 24, 48 and 72 hours after surgery and at ICU discharge, approximately 7 days
  Changes in the metabolomics profile (fold changes) measured by LC-MS and NMR platforms

CONTACTS AND LOCATIONS:
Overall Officials: Nandor Marczin, MD PhD, Study Chair — Imperial College London; Eric EC de Waal, Principal Investigator — UMC Utrecht
Locations (1):
- Harefield Hospital, Harefield, United Kingdom

IPD SHARING:
Plan to Share IPD: No